CLINICAL TRIAL: NCT07221526
Title: SPO2 VALIDATION STUDY - PHILIPS FAST 2025
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-2025-301078-FAST 2025
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: PULSE OXIMETRY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- TEST GROUP 1: Sensor Test Group 1
  * AlarX4 (nasal ala placement)
  * AlarX4 (earlobe placement)
  * M1131AX1
  * M1191BL - As Philips internal silver reference only
  Interventions: Device: NO INTERVENTION
- TEST GROUP 2: Sensor Test Group 2
  * M1133AX5
  * M1133AX6
  * M1191BL - As Philips internal silver reference only
  Interventions: Device: NO INTERVENTION

INTERVENTIONS:
Device: NO INTERVENTION — NO INTERVENTION

SUMMARY:
Clinical investigation is to validate the SpO2 accuracy of the M1133AX5, M1133AX6, and AlarX4 (nasal ala application) SpO2 sensors under test with the Philips FAST Pulse Oximetry technology.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to validate the SpO2 accuracy of the M1133AX5, M1133AX6, and AlarX4 (nasal ala application) SpO2 sensors under test with the Philips FAST Pulse Oximetry technology during non-motion conditions over the range of 70-100% SaO2, when compared with the reference SaO2 obtained from CO-Oximetry analysis of arterial blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Participants accepted into this study must meet all of the following criteria: Participant must have the ability to understand and provide written informed consent
* Participant is an adult between 18-50 years of age
* Participant must be willing and able to comply with study procedures and duration
* Participant is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation (i.e., Raynaud's Syndrome), injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoos (e.g. permanent, Henna) or artificial dyes (e.g. spray tan, artificial tanning lotion) in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the sites utilized.)
* Females who are pregnant
* Females who are trying to get pregnant with confirmation of positive urine pregnancy test
* Participants who have smoked in the last 2 days or participants who have refrained, for at least 48 hours, with COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Participants with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma
  * flu
  * pneumonia / bronchitis
  * shortness of breath / respiratory distress
  * unresolved respiratory or lung surgery
  * emphysema, COPD, lung disease
  * recent COVID with hospitalization
* Participants with self-reported heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * high blood pressure: systolic >140 mmHg or diastolic >90 mmHg on 3 consecutive readings (reviewed during health screen)
  * have had cardiovascular surgery, except successful minor surgery without clinical symptoms (i.e., PFO, PDA) chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
  * implantable active medical device such as pacemaker or automatic defibrillator
* Participants with self-reported health conditions as identified in the Health Assessment Form

  * diabetes
  * uncontrolled thyroid disease
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures)
  * epilepsy
  * history of unexplained syncope
  * recent history of frequent migraine headaches
  * recent symptomatic head injury (within the last 2 months)
  * cancer requiring chemotherapy, radiation, or current treatment
* Participants with known clotting disorders (selfreported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
  * Sickle Cell Trait or Disease
* Participants with self-reported dermatological conditions at sensor application sites

  * severe dermatitis
  * hyperkeratosis
  * nail fungus Participants with severe contact allergies to standard adhesives, latex, silicone or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Participants with severe allergies to iodine (only applicable if iodine is used)
* Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Participants with allergies to ultrasound gel
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio <0.4)
* Unwillingness or inability to remove nail polish, nail jewelry, or artificial nails from test digits. Bruised nail bed of test digits.
* Unwillingness or inability to cut/trim fingernail(s) of test digits if determined length will interfere with correct application of the sensor
* Piercing at application site of the ear or nose sensors that may interfere with correct placement of sensor
* Participants received colored intravascular dye within the past 48 hours (e.g. Indocyanine green, methylene blue, dyes used in cardiac output monitoring)
* Surgical hardware in pathway of Device Under Test
* Other known health conditions should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All
Study Population: The study population will include a minimum of 72 to approximately 90 healthy adult volunteers, divided into 2 test groups.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
SPO2 ACCURACY | OCTOBER 2025-JANUARY 2026
  Accuracy expressed in Arms of SpO2 measurements obtained from the M1133AX5, M1133AX6, and AlarX4 (nasal ala placement) SpO2 sensors under test with the Philips Pulse Oximetry technology over the range of 70-100% SaO2 in comparison to SaO2 as ground truth.

SECONDARY OUTCOMES:
SPO2 ACCURACY | OCTOBER 2025-JANUARY 2026
  Accuracy expressed in Arms of SpO2 measurements obtained from the AlaxX4 SpO2 sensor (earlobe placement) with the Philips Pulse Oximetry technology over the range of 70-100% SaO2 in comparison to SaO2 as ground truth.
DIFFERENTIAL MEAN | OCTOBER 2025-JANUARY 2026
  Maximum differential mean bias as developed by Philips for the M1133AX5, M1133AX6, AlarX4 (nasal ala application), and AlarX4 (earlobe application) in the SaO2 ranges of 70% ≤ SaO2 ≤ 85% and 85% < SaO2 ≤100%.
PIGMENTATION DIFFERENTIAL BIAS | OCTOBER 2025-JANUARY 2026
  Pigmentation differential bias as proposed by ISO for the M1133AX5, M1133AX6, AlarX4 (nasal ala application), and AlarX4 (earlobe application) over the SaO2 range of 80-90%, centered at 85%.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, NP, Principal Investigator — Element Desaturation Lab
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No